CLINICAL TRIAL: NCT03035071
Title: Morbidity In Open Versus Minimally Invasive Hybrid Esophagectomy
Brief Title: Morbidity in Open Versus Minimally Invasive Esophagectomy
Acronym: MIOMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Society Of Surgical Oncology (Other)
Responsible Party: Principal Investigator, Matthias Paireder, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUT-MIOMIE-RCT
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: Minimal-invasive esophagectomy; Esophageal resection; Hybrid esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive esophagectomy (Experimental): minimally invasive (laparoscopic) gastric mobilisation and gastric tube formation.
  Interventions: Procedure: minimally invasive esophagectomy
- open esophagectomy (Active Comparator): open gastric mobilization and gastric tube formation
  Interventions: Procedure: open esophagectomy

INTERVENTIONS:
Procedure: minimally invasive esophagectomy — In the MIE group the laparoscopic procedure was performed for gastric tube formation. The patient was placed in supine position with legs apart. The surgeon stands between the legs using a five-trocar technique. Laparoscopy will be followed by an anterolateral thoracotomy in the fourth intercostal space.
  Arms: minimally invasive esophagectomy
Procedure: open esophagectomy — in the open group the gastric mobilization and gastric tube formation will be perfumed with an open surgical approach. Laparotomy will be performed, followed by an anterolateral thoracotomy in the fourth intercostal space.
  Arms: open esophagectomy

SUMMARY:
The MIOMIE trial is a prospective randomized controlled study comparing open and laparoscopic gastric tube formation in Ivor Lewis esophagectomy. Aim of this trial was to compare the minimally invasive approach with the standard open procedure regarding morbidity and mortality.

DETAILED DESCRIPTION:
Esophageal resection is still associated with considerable morbidity and mortality. Standardized preoperative efforts could increase the outcome of these patients. While early reports of medical pioneers focused particularly on safety and feasibility, more recent studies showed that implementation of minimally invasive esophagectomy (MIE) was widely accepted. Since first reports of MIE, different techniques and adjustments have been discussed. A recent publication of a large prospective trial in Phase II showed the safety of a total minimally invasive approach (video assisted thoracoscopic surgery (VATS) and laparoscopy). Surgical technique however is still a subject of debate and the level of evidence remains still low. Proving feasibility does not warrant a paradigm shift, as experience is an important factor for safety and patient benefit.

The aim of this study was to evaluate morbidity and mortality of open esophagectomy (OE) versus hybrid-MIE in a randomized controlled setting.

Prior to surgery patients will be randomized either the minimally invasive surgery group (laparoscopic gastric tube formation and thoracotomy) or the the open surgery group (open gastric tube formation with an open laparotomy approach). Randomizing tool is the "randomizer" of the medical university of vienna. (link is attached below)

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the esophagus and the esophagogastric junction in (Siewert) type I and II position
* esophageal squamous cell cancer
* patients, who require esophageal resection due to above mentioned diagnosis
* patients, who gave their informed consent

Exclusion Criteria:

* individuals who did not meet the inclusion criteria were excluded from the study.
* patients with tumor localization in the upper third of the esophagus and requiring cervical resection were excluded.
* patients, presenting other than AC or ESCC or showed contraindication for laparoscopy (history of large abdominal surgery or signs of hostile abdomen)
* patients with a history or presence of any other malignancy, except carcinoma in situ or basalioma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2014-11-19 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
morbidity | 30 days
  anastomotic leakage, gastric conduit necrosis and/or pneumonia
mortality | 30 days

SECONDARY OUTCOMES:
ICU stay | 90 days
  length of stay at the intensive care unit (ICU)
hospital stay | 90 days
  length of stay at the hospital
overall survival | 5 years
  long term overall survival
relapse free survival | 5 years
  long term relapse free survival

REFERENCES:
- [Background] Medical Research Council Oesophageal Cancer Working Group. Surgical resection with or without preoperative chemotherapy in oesophageal cancer: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1727-33. doi: 10.1016/S0140-6736(02)08651-8. PMID 12049861
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Low DE, Kunz S, Schembre D, Otero H, Malpass T, Hsi A, Song G, Hinke R, Kozarek RA. Esophagectomy--it's not just about mortality anymore: standardized perioperative clinical pathways improve outcomes in patients with esophageal cancer. J Gastrointest Surg. 2007 Nov;11(11):1395-402; discussion 1402. doi: 10.1007/s11605-007-0265-1. Epub 2007 Aug 31. PMID 17763917
- [Background] Schoppmann SF, Prager G, Langer FB, Riegler FM, Kabon B, Fleischmann E, Zacherl J. Open versus minimally invasive esophagectomy: a single-center case controlled study. Surg Endosc. 2010 Dec;24(12):3044-53. doi: 10.1007/s00464-010-1083-1. Epub 2010 May 13. PMID 20464423
- [Background] Schwameis K, Ba-Ssalamah A, Wrba F, Birner P, Prager G, Hejna M, Schmid R, Asari R, Zacherl J, Schoppmann SF. The implementation of minimally-invasive esophagectomy does not impact short-term outcome in a high-volume center. Anticancer Res. 2013 May;33(5):2085-91. PMID 23645759
- [Background] Messager M, Pasquer A, Duhamel A, Caranhac G, Piessen G, Mariette C; FREGAT working groupFRENCH. Laparoscopic Gastric Mobilization Reduces Postoperative Mortality After Esophageal Cancer Surgery: A French Nationwide Study. Ann Surg. 2015 Nov;262(5):817-22; discussion 822-3. doi: 10.1097/SLA.0000000000001470. PMID 26583671